CLINICAL TRIAL: NCT04149249
Title: CONNECT: Smoking Cessation and Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-25632; NCI-2018-03884 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 186515 (Other: University of California, San Francisco)
Record Dates: First submitted 2019-10-09; First posted 2019-11-04 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Smoking Cessation
Keywords: quitting; smoking; smoking cessation tool; smoking cessation; quit smoking; smoking cessation resources; smoking cessation barriers; smoking cessation intervention tool
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (CONNECT) (Experimental): Patients complete CONNECT, the Video Doctor over 30-45 minutes on an iPad in the waiting room before their lung cancer screening test appointment.
  Interventions: Other: Computer-Assisted Intervention Video Doctor
- Control Group (Active Comparator): Patients complete CONNECT assessment only over 30-45 minutes on an iPad in the waiting room before their lung cancer screening test appointment.
  Individuals who are randomized to the control group will undergo the same assessment questions and all follow up assessments like the intervention group. Instead of viewing and participating in the interactive Video Doctor about Smoking Cessation, they receive a handout containing smoking cessation resources.
  Interventions: Other: Computer-Assisted Intervention no Video Doctor

INTERVENTIONS:
Other: Computer-Assisted Intervention Video Doctor — Complete CONNECT: participants will undergo in-person assessment questions and follow-up assessment questions. They will view and participate in the interactive Video Doctor about Smoking Cessation.
  Arms: Experimental: Intervention Group (CONNECT)
Other: Computer-Assisted Intervention no Video Doctor — Individuals who are randomized to the control group will undergo the same assessment questions and all follow up assessments like the intervention group. Instead of viewing and participating in the interactive Video Doctor about Smoking Cessation, they receive a handout containing smoking cessation resources.
  Arms: Control Group

SUMMARY:
This clinical trial studies the impact of CONNECT on biochemically confirmed smoking abstinence among diverse current smokers who are undergoing lung cancer screening.

DETAILED DESCRIPTION:
The study team will develop and test a novel smoking cessation intervention, CONNECT, which will start at the time an individual is receiving lung cancer screening (LCS). CONNECT will include an interactive Video Doctor which will provide participants with information tailored to their individual responses as well as proactive outreach using brief telephone calls and text messaging to follow up smokers with motivation enhancement to refer and engage patients in evidence based smoking cessation interventions (such as quitline utilization). After development and usability testing, we will conduct a small feasibility study followed by a pilot randomized controlled trial to estimate the impact of CONNECT on biochemically confirmed 30-day smoking abstinence among diverse current smokers seen at the San Francisco Veterans Affairs Medical Center and the University of California San Francisco Division of General Internal Medicine. Participants will be randomized to CONNECT or a control condition. Data will include self-report from participants obtained at baseline, 1 and 3 months, and the electronic health record. Outcomes will be biochemically confirmed 30-day smoking abstinence at 3 months post LCS and satisfaction as well as self-reported quit attempts, and use of evidence-based smoking cessation resources (quitline, pharmacotherapy or counseling). The knowledge gained will provide the pilot data necessary to apply for a larger study to test our novel intervention for promoting smoking cessation among a diverse population of high-risk smokers undergoing Lung Cancer Screening.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-80
* Male or female
* English speaking
* Have an already scheduled low-dose computed tomography (LDCT) visit
* Smoke at least 1 cigarette in the last 7 days
* Have a phone that can receive text messages.

Exclusion Criteria:

* Younger than 55 or older than 80
* Does not speak English
* Does not have a scheduled low-dose computed tomography (LDCT) visit
* Does not smoke at least 1 cigarette in the last 7 days
* Does not have a phone that can receive text messages.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Assessing 30-day smoking abstinence at 3 months post lung cancer screening. | Up to 3 months from date of lung cancer screening appointment.
  Biochemically confirmed 30-day smoking abstinence at 3 months post lung cancer screening.
Number of participants with Self-reported quit attempts | Up to 3 months from date of lung cancer screening appointment.
  Self-reported quit attempts will be measured to assess smoking behavioral changes.
Percentage of participants who used of evidence-based smoking cessation resources | Up to 3 months from date of lung cancer screening appointment.
  Use of evidence-based smoking cessation resources such as quitline, pharmacotherapy or counseling will be measured to assess smoking behavioral changes.

SECONDARY OUTCOMES:
Change in Participation rate over time | Up to 18 months.
  Participation rate, including those who decline to participate and who drop out will be reported as proportions. The data will be compared between the two groups (intervention and control) using the appropriate general linear models with generalized estimating equations (GEE) to account for provider clusters.
Change in intervention component completion rates over time | Up to 18 months.
  Intervention component completion rates, including those who decline to participate and who drop out will be reported as proportions. The data will be compared between the two groups (intervention and control) using the appropriate general linear models with generalized estimating equations (GEE) to account for provider clusters.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Walsh, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsoh JY, Kohn MA, Gerbert B. Promoting smoking cessation in pregnancy with Video Doctor plus provider cueing: a randomized trial. Acta Obstet Gynecol Scand. 2010;89(4):515-523. doi: 10.3109/00016341003678419. PMID 20196678
- [Background] van der Aalst CM, de Koning HJ, van den Bergh KA, Willemsen MC, van Klaveren RJ. The effectiveness of a computer-tailored smoking cessation intervention for participants in lung cancer screening: a randomised controlled trial. Lung Cancer. 2012 May;76(2):204-10. doi: 10.1016/j.lungcan.2011.10.006. Epub 2011 Nov 4. PMID 22054915
- [Background] Clark MM, Cox LS, Jett JR, Patten CA, Schroeder DR, Nirelli LM, Vickers K, Hurt RD, Swensen SJ. Effectiveness of smoking cessation self-help materials in a lung cancer screening population. Lung Cancer. 2004 Apr;44(1):13-21. doi: 10.1016/j.lungcan.2003.10.001. PMID 15013579
- [Background] Marshall HM, Courtney DA, Passmore LH, McCaul EM, Yang IA, Bowman RV, Fong KM. Brief Tailored Smoking Cessation Counseling in a Lung Cancer Screening Population is Feasible: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2016 Jul;18(7):1665-9. doi: 10.1093/ntr/ntw010. Epub 2016 Feb 1. PMID 26834052
- [Background] Ferketich AK, Otterson GA, King M, Hall N, Browning KK, Wewers ME. A pilot test of a combined tobacco dependence treatment and lung cancer screening program. Lung Cancer. 2012 May;76(2):211-5. doi: 10.1016/j.lungcan.2011.10.011. Epub 2011 Nov 15. PMID 22088938